CLINICAL TRIAL: NCT04076748
Title: Evaluation of the Efficacy of Intra-nasal Sufentanil for Analgesia of Vaso-occlusive Crisis in Sickle-cell Adults.
Acronym: DREPSUFINDOL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2017/46
Record Dates: First submitted 2019-08-30; First posted 2019-09-03 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Sickle Cell Crisis
Keywords: analgesia; vaso-occlusive crisis; sufentanil; intra-nasal
MeSH Terms: conditions — Vaso-Occlusive Crises; Agnosia | interventions — Sufentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): * Intra Nasal Sufentanil (50 µg.ml-1): Load dose : 0.3 µg. kg-1, Followed by bolus : 5 µg / 10 minutes with 2 bolus maximum.
  As soon as the venous route and ten minutes after the last administration of sufentanil:
  * Morphine IV: 3 mg / 5 minutes.
  * Objective: numeric rating scale (NRS) ≤ 3/10.
  Interventions: Drug: Sufentanil
- Control (Active Comparator): * EMONO : Given by respiratory administration via a face mask at a rate suitable for patient ventilation (generally at least 9l.min-1), Until a venous route is obtained and without exceeding 30 minutes.
  * Morphine IV: Load dose: 0.1mg. kg-1 as soon as possible; Then bolus: 3mg / 5 minutes.
  * Objective: NRS ≤ 3/10
  Interventions: Drug: EMONO

INTERVENTIONS:
Drug: Sufentanil — The intervention is intranasal Sufentanil adminstration, then IV morphine as soon as possible.
  Arms: Experimental
Drug: EMONO — In the control group, patients will receive EMONO then IV morphine as soon as possible.
  Arms: Control

SUMMARY:
The analgesic treatment for vaso-occlusive crisis (VOC) in sickle-cell patients is an emergency. The reference treatment is morphine, which requires a venous way sometimes difficult to obtain in these patients. Sufentanil intranasal has been shown to be effective in traumatology. The objective is to evaluate, in VOC, the efficacy of intranasal sufentanil relayed by morphine IV compared to the usual protocol, Equimolar Mixture of Oxygen-Nitrous Oxide (EMONO) relayed by morphine intravenous (IV).

DETAILED DESCRIPTION:
Pain of VOC in sickle-cell patients seen in the emergency department (ED) is severe. Analgesia is a therapeutic emergency based on intravenous (IV) morphine titration. However, for technical reasons (patient flow in ED, difficult venous access) this treatment is often delayed. The Equimolar Mixture of Oxygen-Nitrous Oxide (EMONO), an inhaled analgesic administered, makes it possible to temporarily and very partially compensate for the major analgesic defect. Its efficacy in this indication has never been demonstrated; it is less effective than opiates during labour and is associated with a risk of addiction. The intranasal (IN) route is used to administer strong opiates such as sufentanil. Sufentanil IN has been shown to be rapidly effective in traumatology. Its duration of action is similar to that of morphine IV but its duration of action is far too short to completely replace it. Its ideal place would therefore be the initial phase of the management while waiting for a venous approach.

The strategy is to propose an intranasal administration of an opioid (Sufentanil) at the initial management of vaso-occlusive crisis in sickle-cell patients in the ED waiting to a venous route for morphine.

Follow-up of the study will be carried out in the ED with numeric rating scale (NRS) measurement every 5 minutes until patient relief (defined by NRS ≤ 3/10). Once relieved, NRS will be measured every 15 minutes for at least 2 hours. Treatment-related side effects will be systematically investigated up to 4 hours after starting treatment. In particular, the respiratory rate and level of consciousness will be measured, and all side effects will be recorded: nausea, vomiting, dizziness, behavioural disorders, pruritus.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years old;
* Sickle-cell patient.
* Signs of a vaso-occlusive crisis (migratory bone pain, which may occur in the limbs, spine, thorax, pelvis, skull) or crisis known as such by the patient;
* Severe pain (NRS ≥ 6/10) on admission to the ED;
* Registered with the social security scheme or his beneficiaries (except AME)
* Signature of free and informed consen.

Exclusion Criteria:

* Strong opioids received in the previous 6 hours;
* Pregnancy or breastfeeding;
* Woman not menopausal nor sterile without effective contraception (HAS criteria)
* Oxygen saturation below 93%;
* Patients who cannot cooperate because of a State of agitation or a Cognitive impairment
* Unable to communicate;
* Unable to do self-assessment;
* Allergy or intolerance to opiates or nitrous oxide.
* Abuse or addiction to opioids
* Liver insufficiency
* Renal insufficiency
* Severe asthma or chronic obstructive bronchopulmonary disease
* Pulmonary disease necessitating oxygen
* Presence of seriousness signs:

  * All respiratory seriousness signs
  * all neurologic signs or consciousness impairment (coma Glasgow scale under 15)
  * hyperthermia over than 39°C
  * Signs of intolerance of acute anemia
  * Signs of hemodynamic failure
  * Known organ failure (renal insufficiency, pulmonary high blood pressure)
  * A description by the patient of a non usual crisis.
* Current treatment with nasal vasoconstrictors is ongoing
* Head injury with suspicion of high intracranial pressure
* Severe thoracic trauma or decompensated respiratory insufficiency
* Contraindications of intranasal administration:

  * Facial trauma
  * Nose or sinusal surgery in the previous 6 months before inclusion
  * Chronic nose and upper airway alteration (ex. facial malformation)
  * Acute nose and upper airway alteration (ex. Epistaxis, acute respiratory infection, sinusitis).
* Contraindication to nitrous oxide
* Contraindication to morphine
* Patient's refusal to participate in the study.
* Previous inclusion in the study of less than 14 days.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2021-07-20 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients relieved (NRS ≤ 3/10) 30 minutes after starting treatment in each group. | From date of inclusion to 30 minutes after
  This proportion is measured thanks to a numeric rating scale (NRS). The scale define pain intensity, range between 0 and 10, 10 being the worst pain imaginable and 0 the absence of pain. The NRS is measured every 5 minutes until patient relief (defined by NRS ≤ 3/10).

SECONDARY OUTCOMES:
Adverse events occuring until 4 hours after treatment initiation. | From date of inclusion to 4 hours after
  This outcome is defined by the proportion of patients with at least one adverse events during the medical care, until 4 hours after treatment initiation.
Morphine consumption (mg) | from date of inclusion to 60 minutes after
  Assessed morphine consumption after treatment initiation, until 60 minutes.
Morphine consumption (mg) | from date of inclusion to 120 minutes after
  Assessed morphine consumption after treatment initiation, until 120 minutes.
Time to obtain an effective analgesia | through study completion, an average of 4 hours
  Defined an average time to obtain an effective analgesia, after treatment initiation
Time to obtain a venous access | through study completion, an average of 4 hours
  Defined an average time to obtain a venous access, after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Eric FRISON, Dr, Study Chair — USMR
Locations (8):
- France (6):
  - Hopital Pellegrin, Bordeaux
  - Hôpital Louis Mourier, Colombes
  - Gonesse Hospital, Gonesse
  - Hôpital Edouard Herriot, Lyon
  - Hôpital Charles Nicolle, Rouen
  - Hôpital Rangueil, Toulouse
- CH de Cayenne, Cayenne, French Guiana
- CHU Pointe à Pitre, Les Abymes, Guadeloupe

IPD SHARING:
Plan to Share IPD: No